CLINICAL TRIAL: NCT01159145
Title: A Randomised, Single Blind, Two-way Cross-over, Single-centre Study to Assess the Pharmacodynamics (Intragastric pH) and Pharmacokinetics After Repeated Oral Administration of D961H 10 mg and Omeprazole 10 mg in Japanese Healthy Male Subjects
Brief Title: Study to Assess the Pharmacodynamics/Pharmacokinetics After Repeated Dosing of D961H 10 mg and Omeprazole 10 mg in Japanese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: D961HC00009
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Pharmacodynamics Study
Keywords: Healthy volunteer; Japanese males; homo-EM/hetero-EM/PM
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- D961H 10 mg capsule (Experimental): 2 way crossover
  Interventions: Drug: D961H
- Omeprazole 10 mg tablet (Experimental): 2 way crossover
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: D961H — Oral, capsule
  Arms: D961H 10 mg capsule
Drug: Omeprazole — Oral, tablet
  Arms: Omeprazole 10 mg tablet

SUMMARY:
The purpose of this study is to assess the pharmacodynamics (intragastric pH) after repeated oral administration of D961H 10 mg and omeprazole 10 mg in Japanese healthy male subjects who are classified by the genotype of CYP2C19 by the assessment of percentage of time with intragastric pH>4 during 24 hours after dose on day 5.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male subjects between 20 and 45 years of age
* Genotype of CYP2C19 has been known as the volunteer panel data
* H. pylori negative has been known by urea breath test as the volunteer panel data.

Exclusion Criteria:

* Significant clinical illness from the 2 weeks preceding the pre-entry visit to the randomisation, as judged by the investigator(s), eg, acute inflammatory disease which requires medical intervention
* Past or present cardiac, renal, hepatic, neurological or gastrointestinal disease, as judged by the investigator(s), eg, sequelae of myocardial infarction, nephritis, hepatitis and cerebral infarction
* Past or present severe allergic disease, hypersensitivity to food or drugs (except for seasonal hay fever), or allergic symptoms requiring medical intervention (eg, anesthetics used at the intragastric pH measurement)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacodynamics (intragastric pH) after repeated administration of D961H 10 mg and omeprazole 10 mg in Japanese healthy male subjects by the assessment of percentage of time with intragastric pH>4. | A range of 24 hrs

SECONDARY OUTCOMES:
To assess the pharmacodynamics (intragastric pH) after repeated administration of D961H 10 mg and omeprazole 10 mg by the assessment of percentage of time with intragastric pH>3 during 24 hours and 24-hour median intragastric pH. | A range of 24 hrs
To assess the pharmacokinetics after repeated administration of D961H 10 mg and omeprazole 10 mg by the assessment of plasma concentrations and AUCt, AUCt, Css,max, tmax, and t1/2 for D961H and omeprazole after dose on day 5. | A range of 24 hours
To assess the safety and the tolerability after repeated administration of D961H 10 mg and omeprazole 10 mg by the assessment of adverse events, laboratory variables, pulse rate, blood pressure, body temperature and 12-lead ECG | Until last visit, 5-7 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Masataka Date, MD PhD, Study Director — AstraZeneca KK; Ippei Ikushima, MD, PhD, Principal Investigator — AstraZeneca KK
Locations (1):
- Research Site, Tokyo, Tokyo, Japan